CLINICAL TRIAL: NCT02021760
Title: Reduction in Infarct Size by Remote Per-postconditioning in Patients With ST-elevation Myocardial Infarction in Stockholm (RECOND)
Brief Title: Reduction in Infarct Size by Remote Per-postconditioning in Patients With ST-elevation Myocardial Infarction
Acronym: RECOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Pernow (Other)
Responsible Party: Sponsor-Investigator, John Pernow, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECOND
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Ischemic per-postconditioning (Active Comparator): Remote conditioning is induced by inflation of a blood pressure cuff around the left thigh to 200 mmHg or 20 mmHg above systolic blood pressure (if >180 mmHg) for 5 min followed by deflation for 5 min. At least one of these conditioning cycles is performed before PCI is initiated. If time allows, cycles of remote conditioning (5 min leg ischemia and 5 min reperfusion) are repeated until PCI is performed. Following reperfusion, defined as first balloon inflation, four additional cycles of remote conditioning will be performed.
  Interventions: Procedure: Primary Percutaneous Coronary Intervention
- Sham (Sham Comparator): The sham procedures include application of the cuff around the thigh but it is not inflated.
  Otheriwize normal primary PCI.
  Interventions: Procedure: Primary Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Primary Percutaneous Coronary Intervention — Primary Percutanous Coronary Intervention is performed in both Groups.

SUMMARY:
* Trial objective: To test the hypothesis that remote per-postconditioning in connection with primary PCI will reduce myocardial infarct size patients with STEMI.
* Trial Design: Placebo controlled randomized study with parallel groups
* Primary Endpoint: Myocardial infarct size expressed as a percentage of the myocardium at risk determined by Cardiac Magnetic Resonance (CMR) day 4-7
* Efficacy Parameters: Myocardial infarct size expressed as a percentage to the myocardium at risk determined by CMR at 6 months.
* Global left ventricular function determined by left ventricular ejection fraction determined by CMR.
* Microvascular obstruction determined by CMR day 4-7. Quantified ECV (extracellular volume) in left ventricular as myocardium at risk day 4-7 and remodelling parameters day 180.
* Safety Parameters: Major adverse cardiovascular events.

DETAILED DESCRIPTION:
See above. 3 patients left to include.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for primary PCI.
* Chest pain indicating myocardial ischemia with a duration >30 minutes and < 6 hours prior to randomization.
* ST elevations >0.1 mV (>0.2 mV in V2-V3) in > two contiguous leads in V1-V6.
* Informed consent.

Exclusion Criteria:

* Previous myocardial infarction based on medical history or Q-wave on ECG in other area
* Left Bundle Branch Block on ECG.
* Previous CABG
* Cardiac arrest
* Any contraindication for CMR.
* Clinical symptoms of claudication
* Treatment with glibenclamide or cyclosporine on admission.
* Any condition that may interfere with the possibility for the patient to comply with or complete the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size expressed as a percentage of the myocardium at risk determined by Cardiac Magnetic Resonance | 4-7 days following index event

SECONDARY OUTCOMES:
Myocardial infarct size expressed as a percentage to the myocardium at risk determined by Cardiac Magnetic Resonance | 6 months following index event

OTHER OUTCOMES:
Global left ventricular function determined by left ventricular ejection fraction determined by CMR. | 4-7 days and 6 months following index event
Microvascular obstruction determined by CMR | 4-7 days following index event
Quantified ECV (extracellular volume) in left ventricular as myocardium at risk | 4-7 days following index event
Myocardial infarct size by CMR expressed as a percentage to the myocardium at risk determined by Bari or modified Approach Score with coronary angiography. | 5-7 days following index event

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, Professor, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Karolinska University Hospital, Stockholm
  - Danderyds Hospital, Stockholm
  - Södersjukhuset, Stockholm